CLINICAL TRIAL: NCT05237895
Title: Evaluation of Serum Endocan Levels in Patients With Gestational Diabetes
Brief Title: Serum Endocan Levels and Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Elif Yıldız, Principal investigator, Gaziosmanpasa Research and Education Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GaziosmanpaşaTREHi
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Gestational Diabetes; Endocan
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Gestational Diabetes (Other): pregnant women who are at 24-26 weeks of gestational age with positive oral glucose tolerance screening test.
  Interventions: Diagnostic Test: Serum Endocan Levels
- Healty Pregnants (Other): pregnant women who are at 24-26 weeks of gestational age with normal oral glucose tolerance screening test.
  Interventions: Diagnostic Test: Serum Endocan Levels

INTERVENTIONS:
Diagnostic Test: Serum Endocan Levels — Detection of Serum Endocan Levels and detection of possible diagnostic association with gestational diabetes

SUMMARY:
In diabetic patients, serum endocan level has been significantly increased in patients and the levels on the long-term complications are correlated. Based on the Iinformation obtained from these studies, it can be said that there is a strong association between diabetes and serum endocan levels.

DETAILED DESCRIPTION:
It has been shown that endocan level of plasental tissue in gestational diabtes patients is significantly increased when looking at the same week compared with plasenta tissue samples of helathy pregnancy. From the information obtained from these studies, it can be said that there is a strong association between diabetes mellitus and serum endocan levels. investigators aimed to determine the relationship between serum endocan levels and gestational diabetes in the study.

ELIGIBILITY:
Inclusion Criteria:

* being pregnant at 24-26 weeks of gestation
* having oral glucose toleranse screening test
* age between 18-45 years

Exclusion Criteria:

* having in utero mort fetus
* having a previous diagnosis of diabetes
* having a multiple pregnancy
* having a coronary artery disease
* having preeclampcia
* having a pregnancy obtained by assisted reproductive technology
* using cigarette
* using alcohol

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Detection of diagnostic value of serum endocan levels in patient with gestational diabetes | 3 months
  Identifying diagnostic value of serum endocan by comparing serum levels of endocan in groups.

CONTACTS AND LOCATIONS:
Overall Officials: elif yıldız, MD, Principal Investigator — Gaziosmanpasa Research and Education Hospital
Locations (1):
- Gaziosmanpaşa Treh, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No